CLINICAL TRIAL: NCT02117375
Title: EMISEP : Early Spinal Cord Lesions and Late Disability in Relapsing Remitting Multiple Sclerosis Patients
Acronym: EMISEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A00333-42; PHRC/12-07
Record Dates: First submitted 2014-04-10; First posted 2014-04-17 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; spinal cord; MRI; longitudinal study; disability
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with multiple sclerosis (Experimental): 80 patients / clinical Follow-up at M0, M6, M12, M18, M24, M30, M36, M42, M48, M54 and M60 / spinal cord MRI follow-up at M0, M12, M24, M36 and M60 / brain MRI follow-up at M0, M12, M24, M36 and M60
  Interventions: Device: spinal cord MRI follow-up; Other: clinical follow-up; Other: brain MRI follow-up
- Healthy volunteers (Experimental): 20 healthy volunteers (stability of spinal cord imaging) / spinal cord MRI follow-up at M0 and M24
  Interventions: Device: spinal cord MRI follow-up

INTERVENTIONS:
Device: spinal cord MRI follow-up — Evaluation : focal lesions (number, volume, localisation), atrophy, parameters from Diffusion Tensor Imaging and parameters from Magnetization Transfer Ratio
Other: clinical follow-up — Relapses, treatments, global disability,walking performance, upper limbs motor performance, sphincter disturbances and walking difficulty
  Arms: Patients with multiple sclerosis
Other: brain MRI follow-up
  Arms: Patients with multiple sclerosis

SUMMARY:
The purpose of this study is to evaluate the prognostic value of early focal lesions and early diffuse lesions on ambulatory disability progression within 5 years after clinical onset.

DETAILED DESCRIPTION:
Prospective, multicentric study

ELIGIBILITY:
Patients with multiple sclerosis:

Inclusion Criteria:

* Relapsing Remitting Multiple Sclerosis patients (Mac Donald 2010 criteria)
* First clinical event < 1 year
* Brain MRI > 9 lesions or/and spinal cord attack with focal lesion on spinal cord MRI
* Score Expended Disability Status Scale < 3
* Age between 18 and 40 years

Exclusion Criteria:

* Multiple Sclerosis progressive
* Patients treated with immunosuppressive therapy
* Pregnancy

Healthy volunteers:

Inclusion Criteria:

-Age between 18 and 40 years

Exclusion Criteria:

-Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Progressive neurological disability | 5 years
  Measurement by Expended Disability Status Scale

SECONDARY OUTCOMES:
Progressive ambulatory disability | 5 years
  Measurement by the 25-foot timed-Walked test and 6 minutes walking
Progressive disability in the upper limbs | 5 years
  Measurement by the nine-hole peg test
Progressive urinary disability | 5 years
  Measurement by the questionnaire Qualiveen
Progressive difficulty walking | 5 years
  Measurement by the Multiple Sclerosis Walking Scale 12

CONTACTS AND LOCATIONS:
Overall Officials: Gilles GE Edan, Principal Investigator — CHU Rennes; Bruno BB Brochet, Principal Investigator — University Hospital, Bordeaux; Thibault TM Moreau, Principal Investigator — CHU Dijon; Sandra SV Vukusic, Principal Investigator — Hospices civils Lyon; Jean JP Pelletier, Principal Investigator — AP-HM; Marc MD Debouverie, Principal Investigator — CHU NANCY; Bruno BS Stankoff, Principal Investigator — Pitié Salpêtrière; Ayman AT Tourbah, Principal Investigator — CHU REIMS; Jérôme JD De Seze, Principal Investigator — CHU Strasbourg; David DB Brassat, Principal Investigator — University Hospital, Toulouse; Pierre PL Labauge, Principal Investigator — University Hospital, Montpellier; Thibaut TM Moreau, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Rennes, Rennes, France

REFERENCES:
- [Derived] Gros C, De Leener B, Badji A, Maranzano J, Eden D, Dupont SM, Talbott J, Zhuoquiong R, Liu Y, Granberg T, Ouellette R, Tachibana Y, Hori M, Kamiya K, Chougar L, Stawiarz L, Hillert J, Bannier E, Kerbrat A, Edan G, Labauge P, Callot V, Pelletier J, Audoin B, Rasoanandrianina H, Brisset JC, Valsasina P, Rocca MA, Filippi M, Bakshi R, Tauhid S, Prados F, Yiannakas M, Kearney H, Ciccarelli O, Smith S, Treaba CA, Mainero C, Lefeuvre J, Reich DS, Nair G, Auclair V, McLaren DG, Martin AR, Fehlings MG, Vahdat S, Khatibi A, Doyon J, Shepherd T, Charlson E, Narayanan S, Cohen-Adad J. Automatic segmentation of the spinal cord and intramedullary multiple sclerosis lesions with convolutional neural networks. Neuroimage. 2019 Jan 1;184:901-915. doi: 10.1016/j.neuroimage.2018.09.081. Epub 2018 Oct 6. PMID 30300751